CLINICAL TRIAL: NCT01453452
Title: S1008: Feasibility Study of a Physical Activity and Dietary Change Weight Loss Intervention In Breast and Colorectal Cancer Survivors, Phase II
Brief Title: S1008: Exercise, Diet, & Counseling in Improving Weight Loss in Overweight Female Breast or Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S1008; S1008 (Other: SWOG); U10CA037429 (NIH); NCI-2011-03539 (Other: CTRP)
Record Dates: First submitted 2011-10-14; First posted 2011-10-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Anxiety Disorder; Breast Cancer; Cognitive/Functional Effects; Colorectal Cancer; Depression; Fatigue; Pain; Psychosocial Effects of Cancer and Its Treatment; Weight Changes
Keywords: weight changes; fatigue; depression; anxiety disorder; pain; cognitive/functional effects; psychosocial effects of cancer and its treatment; cancer survivor; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Colorectal Neoplasms; Depression; Fatigue; Pain; Body Weight Changes; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise and Lifestyle counseling (Experimental): Patients will receive behavioral dietary intervention & counseling intervention by phone, exercise intervention at Curves(R) facility, and take a quality-of-life assessment online.
  Interventions: Behavioral: behavioral dietary intervention; Behavioral: exercise intervention; Other: counseling intervention; Procedure: quality-of-life assessment

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Reduce caloric intake by 500 kcal/day, increase fruit and vegetable intake to 5 or more servings per day, and limit daily calories from fat to be < 30%. Diet will be measured using 3 repeated 24-hr diet recalls. Participants will receive information on the recommended dietary modifications via mailed materials and telephone counseling sessions.
Behavioral: exercise intervention — 150 min/wk of moderate exercise through use of the Curves® centers, engage in physical activity outside of Curves®, and use pedometers to track activity.
Other: counseling intervention — 14 40-min behavioral counseling sessions via telephone with the goal of increasing intervention adherence and increasing participant retention.
Procedure: quality-of-life assessment — PROMIS-43 - online questionnaire to assess quality of life.

SUMMARY:
RATIONALE: Physical activity, diet, and counseling may help breast and colorectal cancer survivors to lose weight and improve their quality of life.

PURPOSE: This phase II trial studies how well exercise, diet, and counseling work in improving physical activity and weight loss in overweight women who are breast and colorectal cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of a 12-month community-based combined physical activity and dietary change weight-loss intervention in overweight and sedentary female breast and colorectal cancer survivors recruited via the Southwest Oncology Group (SWOG).
* To estimate the effect size of the intervention on weight loss at 12 months.

Secondary

* To measure changes in anthropometric measures from baseline (body mass index [BMI], waist and hip circumference) at 6 and 12 months and body composition (% body fat as assessed by dual-energy X-ray absorptiometry [DXA] scan) at 12 months.
* To measure changes in minutes spent per week in moderate-to-vigorous aerobic activity from baseline using Curves attendance records and a 7-day physical activity assessment at 6 and 12 months.
* To measure changes from baseline to 6 and 12 months in dietary intake of carotenoids via serum carotenoid measures.
* To assess changes from baseline to 6 and 12 months in perceived benefit of dietary change, physical activity, and weight loss after a cancer diagnosis.
* To measure changes from baseline in metabolic and hormonal biomarkers associated with breast and colorectal cancer recurrence risk (fasting insulin, fasting glucose, hemoglobin A1C, bioavailable estradiol, free testosterone, and adiponectin) at 6 and 12 months.
* To assess changes from baseline in anxiety, depression, fatigue, sleep, satisfaction with social roles, pain, and physical function using the PROMISE-43 at 6 and 12 months.
* To assess baseline predictors (medical history, health behaviors, quality of life) of subjects who adhere to and complete the intervention.
* To assess the diversity of subjects who enroll and complete the intervention.
* To assess the availability and acceptability of the Curves fitness centers at 12 months.
* To explore changes in DNA methylation.
* To assess the intervention and study process via open-ended interviews with SWOG sites and Curves franchises.
* To measure changes in anthropometric measures and assess feasibility of extended follow-up at 24 and 36 months.
* To assess the safety of the Curves® fitness centers for this population by assessing self-reported changes in lymphedema and any injuries as measured at 6 and 12 months.

OUTLINE: Participants are stratified according to type of cancer (breast vs colorectal).

Participants are instructed to practice 30-45 minutes of medium-to-hard exercise 5-7 days a week at a Curves fitness center (paid by study) or outside Curves for 12 months. Participants receive written materials on physical activity guidelines for survivors and a pedometer to track their physical activity outside Curves. They also receive the Curves Fitness & Weight Management Plan and are instructed to follow a "higher carbohydrate" diet plan, which promotes a 1,500 kcal/day diet that is high in fruit and vegetables consisting of 30% protein, 45% carbohydrates, and 25% fat. In addition, participants receive the dietary guidelines for cancer survivors, which recommend eating 5 or more servings of fruit/vegetables per day, a diet high in whole grains, low in saturated fat, low in sugary foods, and low in alcohol. Participants receive 14 behavioral-counseling sessions by telephone with the goal to increase intervention adherence and participation retention. Each session lasts 40 minutes and occurs weekly on weeks 1-5 and then every 6 weeks by month 6. Participants receive monthly email newsletters with health tips and motivational messages to encourage adherence and retention to the study program. Counselors also conduct three 24-hour dietary recall assessments and 1 physical activity assessment at 6 and 12 months.

Participants complete a PROMIS-43 quality-of-life questionnaire at 6 and 12 months via internet, mail, or telephone.

Participants also undergo blood sample collection at baseline and at 6 and 12 months for fasting glucose and insulin tests, and biomarker studies. Anthropometric measurements (height, weight, waist, and hip circumference) are also collected.

After completion of study intervention, participants are followed up at 24 and 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participants must be women with a previous diagnosis of stage I, II, or III invasive breast cancer or colorectal cancer

  * Participants must have no evidence of disease at the time of registration and no history of metastases (M0)
* Participants must have a body mass index ≥ 25 kg/m^2 measured within 28 days of registration
* Participants must be considered sedentary (defined as < 60 minutes of moderate to vigorous physical activity per week; moderate exercise defined as exercising to the point of sweating)
* Participants must be willing to submit blood samples for biomarkers (insulin, glucose, HgbA1C, estradiol, and testosterone) and undergo DXA scans, and must be given the option to consent for specimen submission for banking and future translational medicine studies
* Participants must be willing and able to attend a Curves fitness center at least 3 times per week for 12 months

PATIENT CHARACTERISTICS:

* Participants must be post-menopausal, as defined by at least one of the following:

  * At least 12 months since the last menstrual period
  * Prior bilateral oophorectomy
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable) AND follicle-stimulating hormone (FSH) values consistent with the institutional normal values for the post-menopausal state

    * If participant is under the age of 55, FSH levels must be obtained within 28 days prior to registration
* Zubrod performance status of 0
* Participants must have no abnormal changes on a regular (non-nuclear) cardiovascular exercise stress test (using a treadmill or bicycle) as measured by electrocardiogram (EKG)

  * EKG must be within institutional limits of normal
  * Results of previous cardiac exercise stress test may be used as long as it was done within 3 months prior to registration
* Participants must not have evidence of uncontrolled hypertension
* Participants with diabetes, pre-diabetes, and/or metabolic syndrome must have HgbA1C ≤ 8% within the past 28 days

  * Current use of diabetes medications is allowed
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the participant has been disease-free for > 5 years
* Participants must not be active smokers within past 90 days; active smoking is defined as any smoking, even a puff
* Participants must have regular access to the internet in order to receive monthly nutrition-program newsletter e-mails and to complete study questionnaires online
* Participants must be able to understand, speak, and read English
* Participants must have a home phone or cell phone and agree to participate in the 14 (40-minute) behavioral counseling sessions and 9 (20-30-minute) telephone interviews
* Participants must have a baseline physical exam and physician clearance (primary care provider, medical oncologist, or surgical oncologist) to participate in the weight loss and exercise prior to enrollment within 60 days of registration; copy of physician clearance document must be submitted

PRIOR CONCURRENT THERAPY:

* Participants must be 90 days to 730 days post-surgery, chemotherapy, and radiation therapy

  * Current hormonal therapy is allowed among breast cancer participants
  * Other concurrent anti-cancer therapies, including Herceptin, are not allowed
  * Surgery is defined as any major surgical procedure (resection or reconstructive) that would preclude inclusion in the exercise program

    * If the participant has had a remedial surgical procedure (e.g., revision of reconstruction) or persistent complications from her original operation, approval will be obtained from the participant's surgeon prior to enrollment

      * Persistent complications may include, but are not limited to, prolonged wound healing, hernias, or ostomy prolapse

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Attendance of ≥ 2 Curves sessions/week for a minimum of 36 of the 52 weeks of intervention | 1 year from registration
Increase in fruit and vegetable consumption by 1 full serving per day (not including iceberg lettuce, potatoes, or fruit juices) OR reduce caloric intake by 100 kcal/day | 1 year from registration

SECONDARY OUTCOMES:
Changes in anthropometric measures (weight, BMI, waist circumference, hip circumference) | 1 year from registration
Changes in body composition (% body fat as assessed by DXA scan at 12 months only) | 1 year from registration
Changes in minutes spent per week in moderate-to-vigorous intensity aerobic activity using Curves attendance records and a 7-day physical activity recall assessment | 1 year from registration
Changes in dietary intake patterns based on three separate 24-hour diet recalls | 1 year from registration
Changes in metabolic and hormonal biomarkers associated with breast and colorectal cancer-recurrence risk (fasting insulin, fasting glucose, hemoglobin A1C, bioavailable estradiol, free testosterone, and adiponectin) | 3 years
Changes in anxiety, depression, fatigue, sleep, satisfaction with social roles, pain, and physical function as measured by the PROMIS-43 | 1 year from registration
DNA methylation patterns | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, PhD, ND, Study Chair — Herbert Irving Comprehensive Cancer Center; Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (58):
- United States (58):
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Columbia University Medical Center, New York, New York
  - Cancer Centers of the Carolinas - Faris, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville CCOP, Greenville, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Southwest Oncology Group, San Antonio, Texas
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Greenlee H, Lew DL, Hershman DL, Newman VA, Hansen L, Hartman SJ, Korner J, Shi Z, Sardo Molmenti CL, Sayegh A, Fehrenbacher L, Lo S, Klemp J, Rinn K, Robertson JM, Unger J, Gralow J, Albain K, Krouse R, Fabian C. Phase II Feasibility Study of a Weight Loss Intervention in Female Breast and Colorectal Cancer Survivors (SWOG S1008). Obesity (Silver Spring). 2018 Oct;26(10):1539-1549. doi: 10.1002/oby.22269. Epub 2018 Sep 11. PMID 30272836